CLINICAL TRIAL: NCT02588482
Title: Comparison Between High-density Electroencephalography and Conventional Electroencephalography to Diagnose the Presence of Consciousness in Post-anoxic Comatose Patients
Brief Title: Comparison Between High-density Electroencephalography and Conventional Electroencephalography for Comatose Patients
Acronym: COMETIQUE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and feasability issues
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R/2012/46
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Post Anoxic Coma
Keywords: electroencephalography (EEG); mismatch negativity (MMN)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- electroencephalography recording (Experimental): Cerebral measurements from high-density and conventional electroencephalography are recorded simultaneously
  Interventions: Device: high-density electroencephalography; Device: Conventional electroencephalography

INTERVENTIONS:
Device: high-density electroencephalography — Auditory stimulations during electroencephalography recording
Device: Conventional electroencephalography — Auditory stimulations during electroencephalography recording

SUMMARY:
The purpose of this study is to measure whether high-density electroencephalography can improve the detection of electrophysiological signs of awareness compared to conventional electroencephalography in post-anoxic comatose patients

ELIGIBILITY:
Inclusion Criteria:

* post anoxic coma
* over 18 years old
* agreement from families
* alive 4 days after the beginning of coma

Exclusion Criteria:

* traumatic coma
* non-traumatic but not anoxic coma
* patients with severe comorbidity previous to coma
* refusal of families to participate to the study
* contraindication to a high-density electroencephalography exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06-17 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Number of patients who recovered and who presented a mismatch negativity in high-density but not conventional electroencephalography | 4 days after the beginning of coma
  mismatch negativity is an electrophysiological response recorded after the presentation of deviant auditory stimulations Recovery is assessed 1 month after the beginning of coma

SECONDARY OUTCOMES:
Number of patients who recovered and who presented a mismatch negativity in high-density but not conventional electroencephalography | 7 days after the beginning of coma
Number of patients who recovered and who presented a mismatch negativity in high-density but not conventional electroencephalography | 19 days after the beginning of coma

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Moulin, MD, PhD, Principal Investigator — Service de neurologie, CHRU Besançon
Locations (1):
- CHRU Besançon, Besançon, Franche-Comte, France